CLINICAL TRIAL: NCT05437887
Title: Study of the Effects on the Gut Microbiota in the Patients of Atopic Dermatitis Before and After the Treatment of Fucoidan.
Brief Title: Effects of Fucoidan on the Gut Microbiota in the Patients of Atopic Dermatitis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Principal Investigator, YANG SIEN-HUNG, Director of Department of Traditional Chinese Medicine, Chang Gung Memorial Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202200413A3
Record Dates: First submitted 2022-06-14; First posted 2022-06-29 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Atopic Dermatitis
Keywords: atopic dermatitis; Fucoidan; Gut microbiota
MeSH Terms: conditions — Dermatitis, Atopic | interventions — fucoidan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fucoidan (Experimental): All patients are in the experimental group.
  Interventions: Dietary Supplement: Fucoidan

INTERVENTIONS:
Dietary Supplement: Fucoidan — All patients consumed fucoidan.

SUMMARY:
Forty patients with physician-identified atopic dermatitis will be enrolled in the study. All patients must be aged between 6 and 60 years old. All patients consumed fucoidan for 3 months.

DETAILED DESCRIPTION:
Atopic dermatitis is an inflammatory disease with about 6-7% in Taiwan. Its clinical manifestations are repeated rashes and itching of the skin. The patient's skin is stimulated to release inflammatory precursor substances, causing the vascular endothelium to produce adhesion molecules to increase the exudation of inflammatory precursor substances and inflammatory cells to the skin of the lesion; it also triggers the differentiation of Th0 in the skin and blood of the lesion into Th2. Th2 further induced increased serum IgE concentration and increased eosinophilia. At the same time, the non-affected skin will further cultivate more Th2 through leukocytes expressing IgE to enhance the allergic response in the acute phase. Studies show that it is related to the increase of TNF-α. The skin in the chronic phase is mainly manifested by dendritic cells, macrophages, eosinophils, and IL-12. An environment rich in these inflammatory cells and substances allows Th0 to differentiate into Th1 and induces IFN-γ expression, resulting in tissue remodeling, thickening, and desquamation of the epidermis (mossy lesions).

Current treatments for atopic dermatitis include moisturizing agents, antipruritic drugs (such as oral antihistamines), oral and topical steroids, immunomodulators, light therapy, and antibiotic therapy for infections. External use of steroid ointments can easily atrophy the skin and is not recommended for long-term use. Although oral antihistamines can relieve itching, they have the side effect of drowsiness, which can cause an inability to concentrate and trance. In addition, the long-term use of oral steroids has excellent side effects on the endocrine and so on, and it is not suitable for use during infection.

Intestinal bacteria have many effects on the human body, including nutrient absorption, the formation of vitamins and hormones, and the prevention of the formation of pathological colonies. In recent years, the research on the impact of intestinal bacteria on human immune function has become more and more understood. Immunity effects include Segmented filamentous bacteria that promote the differentiation of Th17 and Clostridium spp. that promote the development of regulatory T cells. At the same time, researchers have also found that many diseases, including allergies, asthma, diabetes, obesity, tumors, and neuropathy, may be related to intestinal bacteria. Hothe investigatorsver, whether fucoidan will affect the colony changes in the human gut after taking it has not yet been studied. Our past research discussed that fucoidan could improve atopic dermatitis with immunomodulatory effects, and whether it is related to changes in gut bacteria is unknown.

Purpose:

This study hopes to understand whether improving symptoms in patients with atopic dermatitis by fucoidan is related to intestinal flora change.

Therefore, this prospective trial's results are designed to understand further fucoidan consumption's effect on atopic dermatitis-the effects of gut bacteria in patients.

At the same time, the clinical effect of fucoidan on patients with atopic dermatitis can be tested again.

Specimen collection and testing:

The investigators will get twice stool specimens and blood draw, about 5 c.c. each time, at the beginning and end of the study (at the tthe investigatorslfth the investigatorsek.)

ELIGIBILITY:
Inclusion Criteria:

* Volunteer for study enrollment and sign inform consent
* The age of the patients must be between 6 and 60 years old. Both men and women can participate.
* Symptoms meet the diagnostic criteria of Hanifin and Rajka AD
* The severity of SCORAD (SCORing Atopic Dermatitis) is 25-50 points.

Exclusion Criteria:

* Other eczema-like diseases that are not atopic dermatitis, such as contact dermatitis, seborrheic dermatitis, drug reactions, etc., shall be determined by a dermatologist.
* Associated with other skin diseases that may cause itching, as determined by a dermatologist.
* Have bacterial infection or are using oral or injectable western medicines such as steroids, antibiotics, leukotriene antagonists and other immunosuppressants; as well as using phototherapy, immunotherapy, hyposensitivity therapy; full month.
* Those who cannot cooperate with taking the medicine on time. Those who are unable to cooperate with filling out the questionnaire, drawing blood, and leaving stool samples.
* Those who have a history of allergy to fucoidan or have had adverse reactions and hyperthyroidism.
* Severe organ dysfunction, such as impaired renal and hepatic function at the time of initial diagnosis (including chronic kidney disease stage III, IV, V and AST, ALT ≥ 3 times the upper limit of normal), cirrhosis or heart failure, by clinician determination.
* Uncontrollable mental problems or other serious systemic diseases.
* Pregnant or breastfeeding women and all women of childbearing age who do not agree to take appropriate contraceptive measures.

Ages: 6 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-10-04 (Actual); Primary Completion 2024-03-06 (Estimated); Study Completion 2024-03-06 (Estimated)

PRIMARY OUTCOMES:
collect cecal stool for DNA purification and quantitative PCR for analysis of gut microbiota | Assessment of gut microbiota on Day 0 and 3 month after completing treatment
  Changes in gut bacteria before and after consumption of natural small molecule fucoidan in patients with atopic dermatitis.
  1. Cecal stool DNA purification
  2. Quantification of cecal microbiota by quantitative PCR (qPCR)
  3. V3-V5 16S rRNA amplification

SECONDARY OUTCOMES:
Use SCORAD index to measure the severity and extent of skin rash, itching, and sleep disturbance | Assessment on Day 0 and 3 month after completing treatment
  Evaluation of clinical symptoms such as the severity and extent of skin rash, itching, improvement in quality of life and sleep, and the relationship between the reduction in the use of western medicines and changes in intestinal flora by SCORAD index.
  Subjects were required to return for 3 visits. During these 3 outpatient visits, subjects will be asked questions about atopic dermatitis and photographed and recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Sien-hung Yang, Ph.D., Study Director — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No